CLINICAL TRIAL: NCT03496662
Title: A Phase I/II Study to Evaluate the Tolerability and Efficacy of BMS-813160 (CCR2/5 Inhibitor) With Nivolumab and Gemcitabine and Nab-paclitaxel in Borderline Resectable and Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: BMS-813160 With Nivolumab and Gemcitabine and Nab-paclitaxel in Borderline Resectable and Locally Advanced Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); The Foundation for Barnes-Jewish Hospital (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201806007; 1P50CA196510-01A1 (NIH)
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — BMS-813160; Nivolumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Biopsy

STUDY DESIGN:
Intervention Model Description: Part A: 16 patients will be randomized to 1:1 to control or experimental arm through block randomization without stratification factors. After 8 evaluable patients have been enrolled and treated on the control arm, subsequent patients are enrolled only into the experimental arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A - Experimental Dose Level 0 (Experimental): * BMS-813160 300 mg twice per day
  * Nivolumab 30-minute intravenous (IV) infusion at a flat dose of 480 mg on Day 1 of each 28-day cycle
  * Gemcitabine 30-minute IV infusion 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Nab-paclitaxel 30-40-minute IV infusion 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Post-treatment biopsy at the end of cycle 2
  * Patients who achieve stable disease, a partial response, or complete response after the first 2 cycles of treatment will continue to receive 2 more cycles of treatment followed by a restaging scan. Patients thought to have pseudo-progression will continue to receive treatment for 2 more cyclesore cycles
  Interventions: Drug: BMS-813160; Drug: Nivolumab; Drug: Gemcitabine; Drug: Nab-paclitaxel; Procedure: Biopsy; Procedure: Peripheral blood
- Part A - Control (chemotherapy only) (Active Comparator): * Gemcitabine 30-minute IV infusion 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle Nab-paclitaxel 30-40-minute IV infusion 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Post treatment biopsy at the end of cycle 2
  * Patients who achieve stable disease, a partial response, or complete response after the first 2 cycles of treatment will continue to receive 2 more cycles of treatment followed by a restaging scan. Patients thought to have pseudo-progression will continue to receive treatment for 2 more cycles
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Procedure: Biopsy; Procedure: Peripheral blood
- Part B - Dose expansion (Experimental): * BMS-813160 300 mg twice per day
  * Nivolumab 30-minute IV infusion at a flat dose of 480 mg on Day 1 of each 28-day cycle
  * Gemcitabine 30-minute IV infusion 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Nab-paclitaxel 30-40-minute IV infusion 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Post-treatment biopsy at the end of cycle 2
  * Patients who achieve stable disease, a partial response, or complete response after the first 2 cycles of treatment will continue to receive 2 more cycles of treatment followed by a restaging scan. Patients thought to have pseudo-progression will continue to receive treatment for 2 more cycles
  Interventions: Drug: BMS-813160; Drug: Nivolumab; Drug: Gemcitabine; Drug: Nab-paclitaxel; Procedure: Biopsy; Procedure: Peripheral blood

INTERVENTIONS:
Drug: BMS-813160 — BMS-813160 will be supplied by Bristol Myers Squibb
  Arms: Part A - Experimental Dose Level 0; Part B - Dose expansion
Drug: Nivolumab — Nivolumab will be supplied by Bristol Myers Squibb
  Other Names: Opdivo
  Arms: Part A - Experimental Dose Level 0; Part B - Dose expansion
Drug: Gemcitabine — Gemcitabine will be given as per routine care from commercial supply.
  Other Names: Gemzar
Drug: Nab-paclitaxel — Nab-paclitaxel will be given as per routine care from commercial supply.
  Other Names: Abraxane
Procedure: Biopsy — Pre-treatment, end of cycle 2, end of treatment for patients who progress or otherwise do not go to surgery, and surgery for patients who do go to surgery
Procedure: Peripheral blood — -Cycle 1 Day 1 before treatment begins, after 2 cycles of treatment +/- 3 days of mandatory tumor biopsy, end of treatment for patients who progress or otherwise do not go to surgery, and no more than 24 hours prior to time of surgery (if applicable)

SUMMARY:
The purpose of this research study is to learn more about a new combination of drugs being given to treat pancreatic cancer. The drugs being tested are BMS-813160, nivolumab, gemcitabine, and nab-paclitaxel. The investigators will be looking at both the side effects and the way the disease responds to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or borderline resectable pancreatic ductal adenocarcinoma. Patients with clinical suspicion of pancreatic adenocarcinoma can be enrolled for pre-treatment biopsy, and must be histologically confirmed to have adenocarcinoma before being treated on study. Patients with squamous carcinoma, adenosquamous carcinoma or neuroendocrine tumor will be excluded. Tumor Biopsy can be omitted, if deemed by PI and treatment physician, that it may incur immediate, excessive health risks to patients. This determination (rationale and discussion with PI and treating physician) should be clearly documented in the screening visit notes.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 2,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Hemoglobin ≥ 8.5 g/dL
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN (except participants with Gilbert's Syndrome who must have normal direct bilirubin)
  * AST(SGOT)/ALT(SGPT) ≤ 3 x IULN
  * Serum albumin ≥ 3g/dL
  * Creatinine ≤ 1.5 x IULN OR creatinine clearance ≥ 40 mL/min by Cockcroft-Gault for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use at least two forms of contraception (hormonal, barrier method of birth control, abstinence, and must include barrier method) prior to study entry, for the duration of study participation, and through 5 months (for women) or 7 months (for men) after the last dose of treatment on this study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0) or baseline before administration of study treatment. Participants with toxicities attributed to prior anti-cancer therapy that are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum-based therapy, are permitted to enroll.

Exclusion Criteria:

* Prior exposure to chemotherapy or radiation for the disease to be treated on this trial not allowed.
* Previous malignancies (except non-melanoma skin cancers, and in situ bladder, gastric, colorectal, endometrial, cervical/dysplasia, melanoma, or breast cancers) unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period. Other active malignancy requiring concurrent intervention
* Currently receiving any other investigational agents, or exposure to any investigational drug or placebo within 4 weeks of study treatment
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to BMS-813160, nivolumab, gemcitabine, paclitaxel, nab-paclitaxel, or other agents used in the study.
* Prior exposure to anti-PD-1, anti-PD-L1, CCR2/5, or anti-CTLA4 antibodies.
* Taking immunomodulatory agents (including steroids and NSAIDs). A wash-out period of at least 4 weeks or 5 half-lives, whichever is shorter, is required for patients receiving immunomodulatory agents at the time of enrollment.

Note: daily use of low dose aspirin (e.g. 81 mg PO QD) is not considered an immunomodulatory agent and patients are still eligible for enrollment despite taking such medication at a low dose

* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussing with the Principal Investigator
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study treatment except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted.
* History of allogeneic organ or stem cell transplant.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry and again within 24 hours prior to first treatment.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (by PCR).
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. Anti-retroviral agents are known to have potential adverse pharmacokinetic interactions with nivolumab and/or BMS-813160. IN addition, patients not on anti-retroviral agents, regardless of HIV viral load, are at increased risk of lethal infections with marrow-suppressive therapy including chemotherapy. Testing for HIV must be performed at sites mandated by local requirements.
* Requires continued use of warfarin for anticoagulation and cannot stop warfarin or be safely switched to another anticoagulant.
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease or conditions that could interfere with the swallowing or absorption of study medication or inability to tolerate oral medication.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral anti-bacterial, anti-viral, or anti-fungal therapy ≤ 7 days prior to administration of study medication; immunosuppression; autoimmune conditions; underlying pulmonary disease; or psychiatric illness/social situations that would limit compliance with study requirements.
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
  * QT interval corrected for heart rate using Fridericia's formula (QTcF) prolongation > 480 msec
  * History of other clinically significant heart disease (e.g. cardiomyopathy, congestive heart failure with NYHA functional classification III-IV, pericarditis, significant pericardial effusion, or myocarditis)
* Major surgery within 28 days prior to the first study treatment. Participants must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
* Concurrent use of oral or intravenous medications or food which may interfere with BMS-813160 including any strong inhibitors or inducers of CYP3A4 or P-gp is not allowed. These include but are not limited to Class I antiarrhythmics (eg, quinidine, procainamide, dysopiramide, lidocaine, phenytoin, mexiletine, tocainide, flecainide, propafenone, moricizine), Grapefruit and Seville oranges.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - Experimental Dose Level 0: * BMS-813160 300 mg twice per day
  * Nivolumab 30-minute intravenous (IV) infusion at a flat dose of 480 mg on Day 1 of each 28-day cycle
  * Gemcitabine 30-minute IV infusion 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Nab-paclitaxel 30-40-minute IV infusion 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle
  * Post-treatment biopsy at the end of cycle 2
  * Patients who achieve stable disease, a partial response, or complete response after the first 2 cycles of treatment will continue to receive 2 more cycles of treatment followed by a restaging scan. Patients thought to have pseudo-progression will continue to receive treatment for 2 more cycles
Period: Overall Study
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Started | 7 | 8 | 25
Completed (Completion indicates the participant receiving 4 full cycles of treatment.) | 6 | 8 | 16
Not Completed | 1 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Death | 0 | 0 | 2
Not completed — Noncompliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion | Total
Number analyzed (Participants) | 7 | 8 | 25 | 40
Age, Continuous [Median (Full Range); unit: years] | 71.5 [64 to 78] | 72 [60 to 74] | 68 [48 to 81] | 70 [48 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 8 | 18
  Male | 1 | 4 | 17 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 25 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 6 | 5 | 23 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 25 | 40

OUTCOME MEASURES:

1. Primary Outcome: (Part A Experimental Dose Level 0 Only) Safety of the Combination of BMS-813160 Plus Nivolumab Plus Gemcitabine Plus Nab-paclitaxel as Measured by Frequency, Type, and Severity of Adverse Events
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Time Frame: Through 100 days after completion of treatment (approximately 7.5 months)
Population: -Only participants enrolled in Part A- Experimental Dose Level 0 are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Number analyzed (Participants) | 7 | 0 | 0
Participants
  Grade 1-2 anemia | 6 |  |
  Grade 3 anemia | 1 |  |
  Grade 1-2 leukocytosis | 1 |  |
  Grade 1-2 abdominal pain | 2 |  |
  Grade 1-2 constipation | 3 |  |
  Grade 1-2 diarrhea | 2 |  |
  Grade 3 diarrhea | 1 |  |
  Grade 1-2 hemorrhoids | 1 |  |
  Grade 1-2 mucositis oral | 2 |  |
  Grade 1-2 nausea | 6 |  |
  Grade 4 upper gastrointestinal hemorrhage | 1 |  |
  Grade 1-2 vomiting | 3 |  |
  Grade 1-2 chills | 3 |  |
  Grade 1-2 edema limbs | 5 |  |
  Grade 1-2 fatigue | 3 |  |
  Grade 3 fatigue | 3 |  |
  Grade 1-2 fever | 4 |  |
  Grade 1-2 foot pain | 1 |  |
  Grade 1-2 sweating | 2 |  |
  Grade 1-2 activated partial thromboplastin time prolonged | 1 |  |
  Grade 1-2 alanine aminotransferase increased | 4 |  |
  Grade 3 alanine aminotransferase increased | 2 |  |
  Grade 1-2 alkaline phosphatase increased | 4 |  |
  Grade 3 alkaline phosphatase increased | 1 |  |
  Grade 1-2 aspartate aminotransferase increased | 4 |  |
  Grade 3 aspartate aminotransferase increased | 2 |  |
  Grade 1-2 creatinine increased | 2 |  |
  Grade 1-2 lymphocyte count decreased | 3 |  |
  Grade 3 lymphocyte count decreased | 3 |  |
  Grade 1-2 neutrophil count decreased | 1 |  |
  Grade 3 neutrophil count decreased | 3 |  |
  Grade 4 neutrophil count decreased | 1 |  |
  Grade 1-2 platelet count decreased | 7 |  |
  Grade 1-2 white blood cell decreased | 3 |  |
  Grade 3 white blood cell decreased | 3 |  |
  Grade 1-2 anorexia | 5 |  |
  Grade 1-2 dehydration | 1 |  |
  Grade 1-2 hyperglycemia | 3 |  |
  Grade 3 hyperglycemia | 1 |  |
  Grade 1-2 hypoalbuminemia | 5 |  |
  Grade 1-2 hypocalcemia | 2 |  |
  Grade 1-2 hypoglycemia | 1 |  |
  Grade 1-2 hypokalemia | 3 |  |
  Grade 3 hypokalemia | 1 |  |
  Grade 1-2 hyponatremia | 1 |  |
  Grade 3 hyponatremia | 1 |  |
  Grade 1-2 arthralgia | 2 |  |
  Grade 1-2 back pain | 1 |  |
  Grade 1-2 myalgia | 3 |  |
  Grade 1-2 pain in extremity | 2 |  |
  Grade 1-2 vertigo | 1 |  |
  Grade 1-2 dizziness | 4 |  |
  Grade 1-2 dysgeusia | 1 |  |
  Grade 1-2 headache | 2 |  |
  Grade 1-2 paresthesia | 1 |  |
  Grade 1-2 peripheral sensory neuropathy | 5 |  |
  Grade 1-2 tremor | 2 |  |
  Grade 1-2 depression | 1 |  |
  Grade 1-2 insomnia | 1 |  |
  Grade 1-2 cough | 5 |  |
  Grade 1-2 dyspnea | 1 |  |
  Grade 3 dyspnea | 1 |  |
  Grade 1-2 epistaxis | 4 |  |
  Grade 1-2 hoarseness | 1 |  |
  Grade 1-2 nasal congestion | 1 |  |
  Grade 1-2 pneumonitis | 1 |  |
  Grade 1-2 alopecia | 7 |  |
  Grade 1-2 dermatitis | 1 |  |
  Grade 1-2 discoloration | 2 |  |
  Grade 1-2 nail ridging | 1 |  |
  Grade 1-2 pruritis | 1 |  |
  Grade 1-2 rash maculopapular | 3 |  |
  Grade 1-2 skin hyperpigmentation | 1 |  |
  Grade 1-2 acute kidney injury | 1 |  |
  Grade 1-2 dysuria | 1 |  |
  Grade 1-2 hematuria | 1 |  |
  Grade 1-2 proteinuria | 1 |  |
  Grade 3 cholangitis | 1 |  |
  Grade 1-2 cholecystitis | 1 |  |
  Grade 3 gallbladder obstruction | 1 |  |
  Grade 1-2 hypertension | 1 |  |
  Grade 3 hypertension | 2 |  |
  Grade 1-2 hypotension | 2 |  |
  Grade 1-2 thromboembolic event | 1 |  |
  Grade 1-2 chest swelling | 1 |  |
  Grade 1-2 sinus bradycardia | 2 |  |
  Grade 1-2 vaginal bleeding | 1 |  |
  Grade 1-2 bruising | 1 |  |
  Grade 1-2 infusion related reaction | 1 |  |
  Grade 1-2 wound dehiscence | 1 |  |
  Grade 3 sepsis | 1 |  |
  Grade 1-2 gallbladder infection | 2 |  |
  Grade 1-2 upper respiratory infection | 1 |  |

2. Primary Outcome: (Part B and Part A Experimental Dose Level 0 Only): Objective Response Rate
Description: * Objective response rate (ORR) is defined as number of participants with complete response or partial response.
  * Complete Response (CR): Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Normalization of tumor marker level.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through completion of treatment (approximately 4 months)
Population: Part A - Control participants are not evaluable for this outcome measure. 1 participant enrolled in Part A - Experimental Dose Level 0 is not evaluable for this outcome measure as the participant withdrew prior to the imaging scan. 2 participants enrolled in Part B - Dose expansion were not evaluable for this outcome measure as 1 participant withdrew prior to the imaging scan and 1 participant died prior to the imaging scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Number analyzed (Participants) | 6 | 0 | 23
Participants | 1 |  | 6

3. Secondary Outcome: (Part B and Part A Experimental Dose Level 0 Only): Percentage of Patients Whose Disease Becomes Resectable After Treatment
Time Frame: Completion of treatment (approximately 4 months)
Population: Only participants enrolled to Part A - Experimental Dose Level 0 and Part B - Dose expansion were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Number analyzed (Participants) | 7 | 0 | 25
Participants | 2 |  | 11

4. Secondary Outcome: (Part B and Part A Experimental Dose Level 0 Only): Progression-free Survival (PFS)
Description: * PFS is defined as the days from the date of treatment and death or progression, which occurs first. Patients alive without progression or lost to follow-up are censored at the last follow-up.
  * Progressive disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Through completion of follow-up (median length of follow-up 12.15 months, full range 0.43-44.10 months)
Population: Participants in Part A - control were not evaluable for this outcome measure.
Measure: Mean (Full Range); unit: months
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Number analyzed (Participants) | 7 | 0 | 25
months | 13.69 [4.13 to 35.77] |  | 14.00 [0.43 to 44.10]

5. Secondary Outcome: (Part B and Part A Experimental Dose Level 0 Only): Overall Survival (OS)
Description: OS is defined as days from date of treatment to date of death. Patients alive or lost to follow-up are censored at the last follow-up.
Time Frame: Through completion of follow-up (median length of follow-up 17.63 months, full range 0.43-64.47 months)
Population: Participants in Part A - control were not evaluable for this outcome measure.
Measure: Mean (Full Range); unit: months
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
Number analyzed (Participants) | 7 | 0 | 25
months | 22.55 [6.37 to 64.47] |  | 20.39 [0.43 to 52.43]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until the date of surgery, or 100 days after the last dose of treatment on study if patients did not have surgery [median treatment length was 112 days (full range 14-161 days). All-cause mortality data was collected until completion of follow-up (median length of follow-up 17.63 months, full range 0.43-64.47 months).
Arm/Group | Part A - Experimental Dose Level 0 | Part A - Control (Chemotherapy Only) | Part B - Dose Expansion
All-Cause Mortality (participants affected / at risk) | 5/7 | 4/8 | 21/25
Serious Adverse Events (participants affected / at risk) | 4/7 | 5/8 | 17/25
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Experimental Dose Level 0 (N=7) | Part A - Control (Chemotherapy Only) (N=8) | Part B - Dose Expansion (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Coronary vasospasm (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Fever (General disorders) | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 2 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2
Death due to pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Experimental Dose Level 0 (N=7) | Part A - Control (Chemotherapy Only) (N=8) | Part B - Dose Expansion (N=25)
Anemia (Blood and lymphatic system disorders) | 7 | 4 | 25
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Chest swelling (Cardiac disorders) | 1 | 0 | 0
Prolonged QRS (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 7
Belching (Gastrointestinal disorders) | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 3 | 2 | 11
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 14
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Generalized edema (Gastrointestinal disorders) | 0 | 0 | 3
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 1 | 5
Nausea (Gastrointestinal disorders) | 6 | 1 | 15
Vomiting (Gastrointestinal disorders) | 3 | 1 | 9
Body aches (General disorders) | 0 | 0 | 1
Chills (General disorders) | 3 | 2 | 8
Dry mouth (General disorders) | 0 | 0 | 2
Edema limbs (General disorders) | 5 | 4 | 12
Edema trunk (General disorders) | 0 | 1 | 0
Fall (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 6 | 3 | 20
Fever (General disorders) | 3 | 0 | 10
Foot pain (General disorders) | 1 | 1 | 0
Hand pain (General disorders) | 0 | 0 | 1
Leg pain (General disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Sweating (General disorders) | 2 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gallbladder infection (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1
Thrush (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 4 | 17
Alkaline phosphatase increased (Investigations) | 5 | 1 | 12
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 14
Blood bilirubin increased (Investigations) | 0 | 0 | 3
Creatinine increased (Investigations) | 2 | 0 | 2
Hemoglobin increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 3 | 12
Neutrophil count decreased (Investigations) | 5 | 3 | 11
Platelet count decreased (Investigations) | 7 | 3 | 18
Weight loss (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 6 | 4 | 17
Anorexia (Metabolism and nutrition disorders) | 5 | 2 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 3 | 23
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Port pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spine pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 8
Dysgeusia (Nervous system disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 2 | 1 | 10
Lightheadedness (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 2
Pain in extremity (Nervous system disorders) | 2 | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 3 | 13
Tremor (Nervous system disorders) | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 5
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal hypertension (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Dry nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 4 | 18
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Follicular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 7
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail fungus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Pseudocellulittis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 14
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 0 | 3
Hypotension (Vascular disorders) | 2 | 0 | 3
QT corrected interval prolonged (Vascular disorders) | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (DVT) (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03496662/Prot_SAP_000.pdf